CLINICAL TRIAL: NCT05932173
Title: An Open Label, Single-site, Dose-escalation Study Aiming to Evaluate the Efficacy and Safety of Anti-CD19 CAR-T Manufactured by OlyCAR Platform(OlyCAR-019) in the Treatment of Relapsed/ Refractory(r/r) B-Cell Malignancies
Brief Title: A Study of Novel Anti-CD19 CAR-T in Patients With r/r B-Cell Malignancies
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: 920th Hospital of Joint Logistics Support Force of People's Liberation Army of China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KM-PBC920
Record Dates: First submitted 2023-06-27; First posted 2023-07-06 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-07

CONDITIONS: B-Cell Leukemia; B-Cell Lymphoma; B-cell Tumors
Keywords: B Cell; CAR-T; CD19; Leukemia; Lymphoma
MeSH Terms: conditions — Leukemia, B-Cell; Lymphoma, B-Cell; Leukemia; Lymphoma

STUDY DESIGN:
Intervention Model Description: Patients will receive one of the three doses of 0.5-2*10^6/kg, 3-4*10^6/kg, 5-6*10^6/kg.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- OlyCAR-019 Cell Infusion (Experimental): OlyCAR-019 cell infusion will be administered by vein after short-time manufacture.
  Interventions: Biological: Anti-CD19 Autologous CAR-T Cell Infusion

INTERVENTIONS:
Biological: Anti-CD19 Autologous CAR-T Cell Infusion — Autologous T cells modified with anti-CD19 ScFv expression and manufactured by OlyCAR platform
  Other Names: OlyCAR-019

SUMMARY:
It is a single-center, open-labeled, single-arm, non-randomized, investigator-initiated trial aiming to evaluate the efficacy and safety of anti-CD19 CAR-T manufactured by OlyCAR platform (OlyCAR-019) for CD19+ refractory/relapsed B-Cell malignancies.

DETAILED DESCRIPTION:
OlyCAR is a novel CAR-T manufacturing system which allows to generate clinical-use CAR-T cells in short time. This study is going to evaluate the feasibility of CAR-T manufactured by OlyCAR platform in the treatment of B-Cell malignancies. The OlyCAR-019 cells will be infused by vein. Subjects will be followed for safety and efficacy up to 12 weeks. For those with a durable remission 12 weeks after infusion, the follow-up will last for at least 12 months for disease control.

ELIGIBILITY:
Key Inclusion Criteria:

1. A definite diagnosis of relapsed/refractory B-cell malignancies;
2. Male or female, aged 2-75 years;
3. Confirmed detectable disease；
4. Expected survival time >12 weeks;
5. Eastern cooperative oncology group (ECOG) score is 0-2;
6. Adequate liver , kidney and cardiopulmonary function;
7. Women of childbearing age have negative blood pregnancy test before the start of the trial, and agree to take effective contraceptive measures during the trial until the last follow-up; male subjects with partners of childbearing potential agree to take effective contraceptive measures during the trial until the last follow-up;
8. Willingness to complete the informed consent process and to comply with study procedures and visit schedule.

Key Exclusion Criteria:

1. Presence of other concurrent active malignancy; People with severe mental disorders;
2. History of any of the following genetic disorders, such as Fanconi anemia, Schu-Day syndrome, Gerstmann syndrome, or any other known bone marrow failure syndrome;
3. Acute GVHD of grade II-IV or extensive chronic GVHD;
4. Grade III-IV heart failure or myocardial infarction, cardiac angioplasty or stenting, unstable angina pectoris, or other clinically prominent heart disease within one year prior to enrollment;
5. The presence of any indwelling catheter or drainage (e.g., percutaneous nephrostomy, indwelling catheter, bile drainage, or pleural/peritoneal/pericardial catheter), except for patients who are permitted to use dedicated central venous catheters;
6. Human immunodeficiency virus (HIV) seropositivity; Hepatitis B surface antigen positive or hepatitis B core antibody positive, and HBV-DNA positive; Patients with hepatitis C (HCV-RNA quantitative test results positive); Or the presence of other serious active viral or bacterial infections or uncontrolled systemic fungal infections; Patients with severe history of allergy or allergic constitution;
7. A history of autoimmune diseases (e.g., Crohn's disease, rheumatoid arthritis, systemic lupus erythematosus) leading to end-organ damage or requiring systemic immunosuppressive/systemic disease modulating drugs within the past 2 years; Had or is suffering from interstitial lung disease (e.g., pneumonia, pulmonary fibrosis);
8. Had undergone other clinical trials in the 4 weeks prior to participating in this trial;
9. Poor compliance due to physiological, family, social, geographical and other factors, unable to cooperate with the study protocol and follow-up plan;
10. For patients contraindicated with cyclophosphamide and fludarabine chemotherapy;
11. Subjects requiring systemic corticosteroid therapy (prednisone ≥5mg/ day or equivalent dose of another corticosteroid) or other immunosuppressive agents within 1 month after UCAR-T cell reinfusion, except for adverse events;
12. Receiving donor lymphocyte infusion within 6 weeks before enrollment;
13. Pregnant and lactating women;
14. Subjects with any other condition which the investigator considers unsuitable for inclusion in the study.

Ages: 2 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events(AE) after infusion | Up to 12 months after infusion
  The frequency, severity, and laboratory findings of all adverse events/serious adverse events are included.
MTD | Up to 28 days after infusion
  MTD will be determined based on DLTs observed during the first 28 days of study treatment.

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | Up to 3 months after infusion
  Overall Response Rate (ORR) is defined as the proportion of subjects achieving complete remission(CR) and partial response(PR).
Progression-free survival(PFS) | Up to 3 months after infusion
  Progression-free survival(PFS) refers to the time from cell infusion to the first assessment of tumor progression or death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Sanbin Wang, Professor, Principal Investigator — 920th Hospital of Joint Logistics Support Force of People's Liberation Army of China
Locations (1):
- 920th Hospital of Joint Logistics Support Force of People's Liberation Army of China, Kunming, Yunnan, China